CLINICAL TRIAL: NCT01082809
Title: Phase II Study of Sunitinib as Second-line Treatment in Advanced Biliary Tract Carcinoma: Multicenter, Multinational Study
Brief Title: Sunitinib as Second-line Treatment in Advanced Biliary Tract Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ho Yeong Lim, Samsung Medical center, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02-025
Record Dates: First submitted 2010-01-07; First posted 2010-03-09 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Biliary Tract Adenocarcinoma
Keywords: advanced biliary tract carcinoma; Sunitinib
MeSH Terms: interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (No Intervention): Sunitinib, 37.5 mg orally once daily continuously, comprising a 4-week cycle
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 37.5 mg orally once daily continuously, comprising a 4-week cycle

SUMMARY:
The purpose of this study is to determine whether sunitinib as second-line treatment in advanced biliary tract carcinoma

DETAILED DESCRIPTION:
Phase II study of sunitinib as second-line treatment in advanced biliary tract carcinoma: multicenter, multinational study

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. histologically or cytologically confirmed adenocarcinoma of biliary tract
3. unresectable or metastatic
4. ECOG performance status of 0~2
5. measurable or evaluable lesion per RECIST criteria
6. adequate marrow, hepatic, renal and cardiac functions
7. One prior treatment of cytotoxic chemotherapy (including adjuvant treatment within 12 months)
8. provision of a signed written informed consent

Exclusion Criteria:

1. severe co-morbid illness and/or active infections
2. pregnant or lactating women
3. active CNS metastases not controllable with radiotherapy or corticosteroids
4. known history of hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Time to progression | 12months

SECONDARY OUTCOMES:
Safety profile | 12 months
Response rate | 12 months
Duration of response | 12 months
Overall survival | 12 months
Correlative analyses: EGFR mutational analysis, EGFR immunohistochemical staining, RAS mutational analysis, KIT, PDGFRA, PDGFRB, Beta-Catenin (CTNNB1) mutations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ho yeong Lim, M.D,Ph.D, Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yi JH, Thongprasert S, Lee J, Doval DC, Park SH, Park JO, Park YS, Kang WK, Lim HY. A phase II study of sunitinib as a second-line treatment in advanced biliary tract carcinoma: a multicentre, multinational study. Eur J Cancer. 2012 Jan;48(2):196-201. doi: 10.1016/j.ejca.2011.11.017. Epub 2011 Dec 14. PMID 22176869